CLINICAL TRIAL: NCT05653908
Title: REThinkAcademy: Helping Universities to Effectively Care for the Mental Health of College Students in the Digital Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: REThin Academy
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daily monitoring (Experimental)
  Interventions: Other: StudentMood

INTERVENTIONS:
Other: StudentMood — StudentMood is an app that uses ecological momentary assessment method to asses mood and other mental health corelates. Participants will have to complete the application (the mood wheel, heart rate and other behavioral data as well as standardized scales) daily throughout the entire semester

SUMMARY:
The project aims at monitoring mental health and its mechanism in the student population using a longitudinal design and ecological momentary assessment procedure throughout the first semester of college.

ELIGIBILITY:
Inclusion Criteria:

* student in Babes-Bolyai University in the first year

Exclusion Criteria:

* incapacity of accessing the mobile app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rational and irrational beliefs | baseline, pre-intervention
  Attitudes and Beliefs Scale 2 Abbreviated Version (ABS-2 - AV; Hyland et al. 2014)
Changes in rational and irrational beliefs | immediately after the intervention
  Attitudes and Beliefs Scale 2 Abbreviated Version (ABS-2 - AV; Hyland et al. 2014)
Fluctuation in rational and irrational beliefs | during the intervention
  Attitudes and Beliefs Scale 2 Abbreviated Version (ABS-2 - AV; Hyland et al. 2014)
Mental Health | baseline, pre-intervention
  Mental health- The General Health Questionnaire, 12-item version (GHQ-12)(Goldberg &Williams, 1988)
Changes in Mental Health | immediately after the intervention
  Mental health- The General Health Questionnaire, 12-item version (GHQ-12)(Goldberg &Williams, 1988)
Fluctuation in Mental Health | during the intervention
  Mental health- The General Health Questionnaire, 12-item version (GHQ-12)(Goldberg &Williams, 1988)
Mood disorders | baseline, pre-intervention
  DASS Parkitny, L., & McAuley, J. (2010). The depression anxiety stress scale (DASS). Journal of physiotherapy, 56(3), 204.
Changes in mood disorders | Post-intervention (one week after the intervention)
  DASS Parkitny, L., & McAuley, J. (2010). The depression anxiety stress scale (DASS). Journal of physiotherapy, 56(3), 204.
Fluctuation in mood disorders | during the intervention
  DASS Parkitny, L., & McAuley, J. (2010). The depression anxiety stress scale (DASS). Journal of physiotherapy, 56(3), 204.
Fluctuation in academic stress | during the intervention
  Lin, Y. M., & Chen, F. S. (2009). Academic stress inventory of students at universities and colleges of technology. World Transactions on Engineering and Technology Education, 7(2), 157-162.
Fluctuation in life experiences | during the intervention
  Kohn, P. M., Lafreniere, K., & Gurevich, M. (1990). The inventory of college students' recent life experiences: A decontaminated hassles scale for a special population. Journal of behavioral medicine, 13(6), 619-630.
Fluctuations in emotion regulation | during the intervention
  Garnefski, Nadia, and Vivian Kraaij. "Cognitive emotion regulation questionnaire-development of a short 18-item version (CERQ-short)." Personality and individual differences 41.6 (2006): 1045-1053.
Fluctuations in college student stress | during the intervention
  Feldt, R. C. (2008). Development of a brief measure of college stress: The college student stress scale. Psychological reports, 102(3), 855-860.
Fluctuations in stress coping styles | during the intervention
  Lin, Y. M., & Chen, F. S. (2010). A stress coping style inventory of students at universities and colleges of technology. World Transactions on Engineering and Technology Education, 8(1), 67-72.
Student adaptation to college | during the intervention
  College Adaptation Questionaire is a scale ) to assess how well students have adjusted to university life, is a self-report instrument consisting of 18 statements. Respondents indicate on a seven-point rating scale how well each statement applies Van Rooijen, L. (1986). Advanced students' adaptation to college. Higher Education, 15(3), 197-209.

SECONDARY OUTCOMES:
Trauma | baseline, pre-intervention
  Childhood Trauma Screener Witt, A., Öz, Y., Sachser, C. et al. Validation and standardization of the Childhood Trauma Screener (CTS) in the general population. Child Adolesc Psychiatry Ment Health 16, 73 (2022). https://doi.org/10.1186/s13034-022-00506-6
Loneliness | baseline, pre-intervention
  Snape, D., & Martin, G. (2018). Measuring loneliness: guidance for use of the National indicators on surveys. Office for National Statistics.
Fluctuation in loneliness | during the intervention
  Snape, D., & Martin, G. (2018). Measuring loneliness: guidance for use of the National indicators on surveys. Office for National Statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No